CLINICAL TRIAL: NCT01350739
Title: Comparative, Randomized, Open-label Study: Different Incisions to Access the Abdominal Cavity Within the Umbilicus
Brief Title: The Umbilical Access in Laparoscopic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Dauser, MD, MD, St John of God Hospital, Vienna
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Umb11
Record Dates: First submitted 2011-05-08; First posted 2011-05-10 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Scars; Patient Satisfaction; Cosmesis
MeSH Terms: conditions — Cicatrix; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraumbilical incision (Other): an intraumbilical vertical incision is made
  Interventions: Procedure: intraumbilical incision
- infraumbilical incision (Other): incision is done in circular fashion at the inferior boarder of umbilicus
  Interventions: Procedure: infraumbilical incision

INTERVENTIONS:
Procedure: intraumbilical incision — vertical, intraumbilical incision
  Arms: intraumbilical incision
Procedure: infraumbilical incision — incision at the inferior boarder of the umbilicus, circular
  Arms: infraumbilical incision

SUMMARY:
The aim of this study is to access to the abdominal cavity using different incision-types within the umbilical area.

Effects of different incisions on scarring and on the umbilical form will be investigated.

ELIGIBILITY:
Inclusion Criteria:

- patient undergoing laparoscopic surgery

Exclusion Criteria:

* pregnancy
* patients following open abdominal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Scarring related to different accesses at the umbilicus | 3, 12 months
  Appearance of scars will be assessed by means of the Manchester Scar Scale (MSS)

SECONDARY OUTCOMES:
Patient satisfaction with scars | 3, 12 months
  Appearance of the umbilical postoperatively and patient satisfaction with the operative results will be assessed by means of a Body Image Questionnaire (BIQ)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Dauser, MD, Principal Investigator — St John of God Hospital, Vienna
Locations (1):
- Department of Surgery, St John of God Hospital, Vienna, Vienna, Austria